CLINICAL TRIAL: NCT01501396
Title: Treatment of Cancer Anorexia-cachexia Syndrome (CACS) With Mirtazapine and Megestrol Acetate
Brief Title: Megestrol Acetate With or Without Mirtazapine in Treating Cancer Patients With Weight Loss or Loss of Appetite
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 201202023
Record Dates: First submitted 2011-12-20; First posted 2011-12-29 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Anorexia
MeSH Terms: conditions — Anorexia | interventions — Megestrol Acetate; Mirtazapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (megestrol alone) (Experimental): Megestrol acetate 800 mg PO daily x 8 weeks
  Interventions: Drug: Megestrol Acetate
- Arm B (megestrol plus mirtazapine) (Experimental): Megestrol acetate 800 mg PO daily x 8 weeks
  Mirtazapine 15 mg PO at bedtime x 1 week followed by 30 mg PO at bedtime x 7 weeks
  Interventions: Drug: Megestrol Acetate; Drug: Mirtazapine

INTERVENTIONS:
Drug: Megestrol Acetate
  Other Names: BDH 1298; Maygace; Megace; Megestil; Niagestin; Pallace
Drug: Mirtazapine
  Other Names: Remeron
  Arms: Arm B (megestrol plus mirtazapine)

SUMMARY:
This randomized phase II trial studies the safety and efficacy of megestrol acetate given with or without mirtazapine in treating cancer patients with weight loss and loss of appetite. To date, no pharmacologic interventions have been approved by FDA to treat cancer anorexia-cachexia syndrome (CACS). Megestrol acetate has been shown to increase appetite in cancer patients. Adding mirtazapine may provide a much more effective treatment and help improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a histologically or cytologically confirmed solid malignancy
* Patient must be >=18 years old.
* Patient must have shown unintentional weight loss of >= 5% in 6 weeks dating back from time of consent or >= 10% in 6 months dating back from time of consent
* Patient must have a poor appetite (defined as a score of =< 14 on the Simplified Nutritional Appetite Questionnaire (SNAQ)
* Prior diagnostic or therapeutic surgery is allowed as long as the wound has fully healed, the patient has fully recovered from the procedure, and at least 4 weeks have elapsed from the procedure; for needle or core biopsy, or minimally invasive procedures such as chest tube placement, this 4-week recovery period does not apply, but the patient must have recovered fully from the procedure
* Concomitant administration of chemotherapy is permitted but not required
* Prior radiation therapy is allowed for local symptom palliation prior to the start of treatment as long as at least 2 weeks have elapsed from the procedure and the patient has fully recovered from treatment-related toxicities
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Patient must have normal organ and marrow function as defined below:
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Patient must be able to understand and willing to sign a written informed consent document

Exclusion Criteria:

* Patient must not be receiving any other investigational agents
* Patient must not be receiving any tube feeds or parenteral nutrition
* Patient must not be taking either MA or MRZ within 4 weeks prior to enrolling on the study, prior use of either MA or MRZ more than 4 weeks before enrollment is allowed
* Patient must not be taking any medication for appetite stimulation within 4 weeks prior to enrolling on the study; prior use of an appetite stimulant more than 4 weeks before enrollment is allowed
* Patient must not have a known seizure disorder
* Patient must not have received abdominal radiation within 4 weeks of enrolling on the study; patients who have received abdominal radiation more than 4 weeks prior to enrollment may participate in the study, as long as they have recovered from toxicities of radiation therapy
* Patient must not be taking chronic systemic corticosteroids (e.g., prednisone, dexamethasone) within the 4 weeks prior to study entry or while on study (unless as pre-medication for chemotherapy)
* Patient must not have moderate to severe depression defined as score of >= 20 on the Center for Epidemiologic Studies Depression Scale (CES-D)
* Patient must not be taking any anti-depressant therapy within the 4 weeks prior to study entry
* Patient must not be on antipsychotic therapy such as risperidone, quetiapine, clozapine, phenothiazine, or butyrophenone for 30 days prior to study; patient may receive prochlorperazine or other phenothiazines as antiemetic therapy
* Patient must not have a history of phenylketonuria (MRZ compounds contain phenylalanine)
* Patient must not have active dysphagia or gastrointestinal tract obstruction
* Patient must not have a previous history of deep venous thrombosis, pulmonary embolism, or thrombophlebitis
* Patient must not be receiving any other agent to increase appetite or weight such as growth hormone (GH), insulin-like growth factor (IGF-1), growth hormone-releasing hormone, insulin-like growth factor binding protein-3 (IGFBP-3), or cannabinoids within the 6 weeks prior to study entry
* Patient must not have a body mass index (BMI) > 30
* Patient must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to MA or MRZ
* Patient must not have any uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Mirtazapine can cause non-teratogenic adverse effects on the developing human fetus at the recommended therapeutic dose; for this reason and because MA as well as other therapeutic agents used in this trial are known to be teratogenic, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; women of childbearing potential must have a negative pregnancy test prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Response rates for weight gain | Baseline to 8 weeks
  Determine the rates of >= 5% weight gain in the treatment groups. Compare the difference of the response rate between the 2 groups.

SECONDARY OUTCOMES:
Safety and tolerability of MA alone and MA + MRZ | Baseline to 12 weeks (30 days after end of study)
  NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.
Weight change (in lbs) | Baseline to 8 weeks
  Change over time as well as the difference between groups for weight (in lbs) will be analyzed.
Appetite stimulation | Baseline to 8 weeks
  Assessed using Simplified Nutritional Appetite Questionnaire (SNAQ). The change over time as well as the difference between groups will be analyzed.
Quality of life | Baseline to 8 weeks
  Assessed using the Functional Assessment of Anorexia/Cachexia Therapy (FAACT). The Change over time as well as the difference between groups will be analyzed.
Mood assessments | Baseline to 8 weeks
  Measured using CES-D. The Change over time as well as the difference between groups will be analyzed.
Evaluation of biochemical markers | Baseline to 8 weeks
  Explore the relationship between weight gain and serum markers of nutritional status (prealbumin, transferrin, C-reactive protein, TNF-alpha, and IL-1 and IL-6).

CONTACTS AND LOCATIONS:
Overall Officials: Saiama Waqar, M.D., Principal Investigator — Washington University School of Medicine

REFERENCES:
- [Derived] Vita G, Compri B, Matcham F, Barbui C, Ostuzzi G. Antidepressants for the treatment of depression in people with cancer. Cochrane Database Syst Rev. 2023 Mar 31;3(3):CD011006. doi: 10.1002/14651858.CD011006.pub4. PMID 36999619
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu